CLINICAL TRIAL: NCT04358640
Title: Anxiety and Work Resilience Among Tertiary University Hospital Workers During the COVID-19 Outbreak: An Online Survey
Acronym: PSY_CO_CHU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL COVID 2019/JYL-01)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Critical Illness; Sars-CoV2; SARS Pneumonia; Coronavirus Infection; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Critical Illness; Coronavirus Infections; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Employees of Nîmes University Hospital (France): Employees of Nîmes University Hospital (France)

SUMMARY:
For limiting COVID-19 spreading, the World Health Organisation (WHO) recommended worldwide confinement on 2010. In France, unessential institutions were closed on March 14th and population confinement was decided on March 17th.

Quarantine and/or confinement could lead to psychological effects such as confusion, suicide ideation, post-traumatic stress symptoms or anger COVID-19 outbreak highlighted a considerable proportion of health care workers (HCW) with depression, insomnia, anxiety and distress symptoms. In front line, facing the virus with the fear of contracting it and contaminate their closest. During previous outbreaks (H1N1, SARS), HCWs have been shown to experience such negative psychological effects of confinement as well as work avoidance behaviour and physical interaction reduction with infected patients (4-7).

In France, Covid 19 outbeak led to increase ICU bed capacity with a full reorganization of the human resources. Some caregivers were reassigned to newly setup units admitting or not Covid-19 patients. In the same time, non-caregivers were also encouraged to work at home whenever possible. Thus, every hospital staff member's private and professional life could be altered by the Covid-19 outbreak.

As all these changes in the daily life could induce psychological disturbances, the present study was aimed at assessing the acute anxiety level (main objective) of the staff in our Tertiary University Hospital, (6300 employees). Secondarily, the self-reported insomnia, pain, catastrophism and work avoidance behaviour levels were assessed

ELIGIBILITY:
Inclusion Criteria:

* Employees of CHU Nîmes during COVID-19 pandemic
* Approved to participate

Exclusion Criteria:

• Participation refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All employees of ICHU Nîmes participating to the present study will be sent a questionnaire for assessing the potential occurrence of anxiety This evaluation will be performed after the beginning of the outbreak (15 to 45 days)
Sampling Method: Non-Probability Sample
Enrollment: 1784 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Anxiety | 15 to 45 days after the beginning of the outbreak
  Mesured by STAY Scale

SECONDARY OUTCOMES:
Insomnia | 15 to 45 days after the beginning of the outbreak
  Participant suffering of Insomnia
Catastrophism | 15 to 45 days after the beginning of the outbreak
  Participant suffering of catastrophism

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive care unit CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714